CLINICAL TRIAL: NCT03552042
Title: Ageing as a Mindset: A Counterclockwise Experiment to Rejuvenate Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Francesco Pagnini, Assistant Professor of Clinical Psychology, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ageing01
Record Dates: First submitted 2018-05-10; First posted 2018-06-11 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Counterclockwise Program (Experimental): Subjects will participate in an 6-day Counterclockwise Retreat in a retrofitted physical environment circa 1989, which helps the participant psychologically return to a time before diagnosis to re-experience their younger self. Groups will be composed of 10-12 participants plus 3 research assistants/facilitators. Participants will live during the week as if they were in 1989, talking about 1989 events as if they were in the present, and avoiding talking about post-1989 events. Everybody will be invited to participate in conversations and discussions about 1989 in the present tense (presente). Furniture, posters, music, television, newspapers, and technological instruments will all reflect what was available in 1989. Participants will be told not merely to reminisce about this earlier era, but to "inhabit" life in that era, making a psychological leap to be the person they were at the end of the 1980s.
  Interventions: Behavioral: Counterclockwise program
- Active control group (Active Comparator): Participants in the active control group will follow the same agenda of the Counterclockwise Program group, without the constant reference to 1989. The intervention will take place in the same location of the Counterclockwise Program, without any specific change. Activities will mirror the ones of Counterclockwise Program, but participants will not live as if they were younger. The agenda will be the same, but no mention to 1989 will be done. All discussion activities will refer to present days (e.g., instead of discussing the open of the Berlin Wall, they can discuss Brexit or Trump presidency).
  Interventions: Behavioral: Active control group
- No-treatment control group (No Intervention): Non-treated participants will be assessed with the same timeline followed by the other groups. Participants will receive three coupons, for each assessment after the baseline (at T2, T3, and T4) for a two-night break in a location of their choice (among a selection of commercial services).

INTERVENTIONS:
Behavioral: Counterclockwise program — A group of older adults (aged 75+) will take part of a residential role-play game, in which they will relive their previous self, acting as if they were in the year 1989. The whole residential program, which will last one week, is designed to enhance this perception, including a retrofitted environment and social activities that will prime participants to relive that period.
  Arms: Counterclockwise Program
Behavioral: Active control group — Participants in the active control group will follow the same agenda of the Counterclockwise Program group, without the constant reference to 1989. The intervention will take place in the same location of the Counterclockwise Program, without any specific change. Activities will mirror the ones of Counterclockwise Program, but participants will not live as if they were younger. The agenda will be the same, but no mention to 1989 will be done. All discussion activities will refer to present days (e.g., instead of discussing the open of the Berlin Wall, they can discuss Brexit or Trump presidency).
  Arms: Active control group

SUMMARY:
Ageing is generally perceived as a biologically-determined process. There is growing literature, however, that discusses the role of psychological factors in the ageing process. In particular, age-related stereotypes, which reflect the images that people have about the ageing process, seem to have a strong influence on health and life satisfaction, through self-fulfilling prophecy mechanisms. According to the stereotype embodiment theory, mindful changes in these images will promote a change in both the mind and the body, resulting, for example, in a rejuvenation and in a higher quality of life.

The project aims to investigate whether changes in mindsets (i.e., addressing one's age-related stereotypes) can change the ageing process. The psychological components of ageing, as well as how these could be reverted, will be investigated. In other words, the study aims to provide a first answer to the question: "can the mind be used to become younger?" To answer this question, the project will test the efficacy of an intervention labeled "counterclockwise", based on an original, yet un-replicated, pilot study by Ellen Langer, at Harvard. A group of older adults (aged 75+) will take part of a residential role-play game, in which they will relive their previous self, acting as if they were in the year 1989. The whole residential program, which will last one week, is designed to enhance this perception, including a retrofitted environment and social activities that will prime participants to relive that period.

The counterclockwise intervention will be tested against an active control group and a no-treatment group, with a randomized controlled trial. People in the active control group will spend a week in the same location of the counterclockwise intervention, mirroring the same activities, without any kind of time manipulation. Participants in the no-treatment group will only receive the assessment. Ninety participants will be randomly allocated to one of these three groups. Every participant will be assessed for medical, cognitive, psychological, and age appearance, four times: at the recruitment, after the intervention (i.e., after a week for the no-treatment group), and again after 6 and 12 months.

Expected results will be able to promote a mindset-shift not only in the participants but in the general population. The communication plan, which is integrated into the project plan, includes the presentation of the results to communities and associations of older adults, using the experiment as a proof of concept. It will demonstrate that challenging rigid, culturally driven, age-related stereotypes can result in health and well-being improvement. This is expected to lead to a significant improvement of empowerment and perceived control, with the potential to become viral in social communications.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* Cognitively preserved, assessed with a Mini Mental State Examination (Folstein, Robins, & Helzer, 1983) score > 18
* Able to commit the time requested to join the retreat (one full week)
* Live in Milan (Italy), or close enough to travel to attend the assessments

Exclusion Criteria:

* Major disability that involves the use of a wheelchair or technological devices (e.g., communication device, invasive or non-invasive ventilation)
* Recent (<9 months) traumatic events (e.g., death of a close relative, life-threatening events)
* Traumatic events toward the end of the '80s or the beginning of the '90s

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the Short Physical Performance Battery | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Physical function will be assessed with the Short Physical Performance Battery (SPPB), a well-established measure of physical function in older adults (Guralnik et al., 1994). It assesses strength, gait, and balance by examining, respectively: (1) time to rise from a chair and return to the seated position five times; (2) time to walk eight feet; and (3) ability to stand with feet together in the side-by-side, semi-tandem, and tandem positions for 10 seconds. Possible scores ranged from 0 to 12, with a higher score indicating better physical performance. Older individuals who receive lower scores on this measure has increased risk of disability, nursing-home placement, and mortality (Levy, et al., 2014; Guralnik et al., 1994).

SECONDARY OUTCOMES:
Heart rate | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Heart rate (HR) will be assessed with a Nonin 2500C-UNIV Universal Charger for 2500 Series with a mercury palm-style tat us.
Blood pressure | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Blood pressure (BP) will be measured with three 45-second readings on the participant's left harm.
Oxygen saturation | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Oxygen saturation is a term referring to the fraction of oxygen-saturated hemoglobin relative to total hemoglobin in the blood, and it will be measured with a Nonin 2500C-UNIV Universal Charger for 2500 Series.
Respiratory rate | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Respiratory Rate (RR) is the number of breaths per minute, which will be collected to determine whether the respirations are normal, abnormally fast, abnormally slow, or nonexistent.
Memory | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Memory will be assessed with the Babcock Story Recall Test (Freides and Avery, 1991). In this verbal memory test, a brief news is presented, and immediate recall is obtained. The story is then presented a second time, and after administration of intervening tasks, delayed recall is obtained. Scores for several normative samples have been reported and it is considered a valid method for assessing verbal memory. Good inter-rater reliability has previously been reported (Freides & Avery, 1991).
Attentive function | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Attentive function will be evaluated with the Dual Task Performance, a pencil-and-paper test of divided attention, which consists of two components, a digit span task and a visuo-spatial tracking task. Each task is performed both separately and concurrently (Della Sala, et al., 2010).
Psychological well-being | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  The Psychological General Well-being Index (PGWBI) is a questionnaire that assesses well-being. It is composed by 22 items representing six dimensions: anxiety, depressed mood, positive well-being, self- control, general health, and vitality. It is a widely used tool to asses quality of life, and it has excellent psychometric validity (Ruini, C., et al., 2003). The total score ranges from 0 to 110, with higher values indicating higher well-being. Subscale score ranges are: anxiety, 0-25; depressed mood, 0-15; positive well-being, 0-20; self-control, 0-15; general health, 0-15; and vitality, 0-20. Higher scores are associated with better outcomes (i.e., always "positive"). The total score is provided by the sum of the subscales.
Anxiety | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Anxiety will be evaluated with the Geriatric Anxiety Inventory (GAI; Pachana et al., 2007), a 20-item measure of anxiety symptoms, specifically developed for older adults. It has been shown to have adequate internal consistency, test-retest reliability and concurrent validity (Pachana, et al., 2007). The scale ranges from 0 to 60, with higher scores indicating higher levels of anxiety.
Depression | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Depression will be assessed with the Geriatric Depression Scale (GDS; Yesavage et al., 1983), a 30-item self- report measure of depressive symptoms, developed for older adults. The validity and reliability of this tool have been supported through both clinical practice and research (Yesavage et al., 1983). Questions are answered "yes" or "no." One point is assigned to each answer and the cumulative score is rated on a scoring grid, which sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed". The total score ranges from 0 to 30.
Ageing stereotypes | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Ageing stereotypes will be evaluated with the open-ended Image-of-Aging question: "What are the first five words or phrases that come to mind when you think of an older person?" (Levy & Langer, 1994). Three independent raters will score responses on a Likert scale ranging from 1 (very negative) to 5 (very positive), which will be combined as an average, providing one single score. This measure produces responses rated as stereotypical of old age (Levy, Slade, & Gill, 2006), predicts physical recovery (Levy, Slade, Murphy & Gill, 2012), and shows expected variability and cross-cultural patterns (Levy & Langer, 1994).
Appearance | Assessed at recruitment; after completing the intervention, i.e., one week after recruitment for the non-treated control group; at a 6-month follow-up; at a 12-month follow-up
  Participants will be photographed at each assessment to evaluate age appearance. The photos will have a neutral (i.e., white) background and will have the same instructions: "please, smile to the camera". University students will blindly guess the age of every person in each picture. Pictures will be showed online with a random allocation through the Qualtrics suite to at least 200 undergraduate students. The final score for each picture will be the average age guessed by students.

CONTACTS AND LOCATIONS:
Locations (1):
- Università Cattolica del Sacro Cuore, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pagnini F, Cavalera C, Volpato E, Comazzi B, Vailati Riboni F, Valota C, Bercovitz K, Molinari E, Banfi P, Phillips D, Langer E. Ageing as a mindset: a study protocol to rejuvenate older adults with a counterclockwise psychological intervention. BMJ Open. 2019 Jul 9;9(7):e030411. doi: 10.1136/bmjopen-2019-030411. PMID 31289097